CLINICAL TRIAL: NCT07166978
Title: Improving Autistic Children's Experiences of Dental Care With Class-integrated Social Story: a Randomised Controlled Trial and Cost-benefit Analysis
Brief Title: Improving Autistic Children's Experiences of Dental Care With Class-integrated Social Story
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UW24-535
Record Dates: First submitted 2024-11-10; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2024-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive a validated social story ECOHC and reinforcement sessions after baseline recruitment. The developed and validated social story will be distributed to the participants in the intervention group. The same research assistant will visit their SCCCs 8 times to provide weekly class-integrated social story reinforcement sessions at 1-2 months.
  All children will receive dental examinations at their respective SCCCs at 3, 6, 12, 18 months.
  Interventions: Behavioral: Social story
- Control (No Intervention): The control group will not receive any social story or reinforcement session throughout the study period.
  All children will receive dental examinations at their respective SCCCs at 3, 6, 12, 18 months.

INTERVENTIONS:
Behavioral: Social story — Social story is a training method constituting of short stories to convey information in a step-by-step manner, so that ASD children can understand what to expect and how to behave in different situations in daily lives. Social stories have been implemented to introduce dentistry and improve oral hygiene to individuals diagnosed with ASD with promising results. However, the certainty of evidence for its effectiveness in reducing dental fear during dental visit was low as the results were derived from small-scaled non-randomized controlled studies.
  Arms: Intervention

SUMMARY:
Children with autism spectrum disorder (ASD) are more likely to have unmet dental needs. Due to hypersensitivity and oral defensiveness, new or unexpected stimuli during dental examinations often precipitate anxiety and stress. These dental barriers often exacerate the difficulties in managing ASD children during periodic comprehensive dental reviews, which are essential for prevention, early identification and management of oral problems, and maintenance of good oral health.

Social story is a training approach constituting short stories and visual cues designed to convey information in a step-by-step manner, to help ASD children know what to expect and how to behave in different situations in daily life, and to gradually allow them to adjust to essential daily tasks. Our previous publications reported the success of social stories in improving oral health among ASD children, but its use in improving their experience in dental care and reducing their dental fear were only been validated in small-scale trials.

Our team has developed and validated a dental-visit social story (DVSS) in collaboration with a review panel comprising of paediatric dentist, clinical psychiatrist and psychologist, speech and hearing therapist, dental practitioner, occupational therapist, social worker, and caregivers and teachers of ASD preschool children. A randomised controlled trial is conducted to compare and evaluate the clinical efficacy and cost benefits of DVSS among ASD preschool children. ASD preschool children are recruited and randomly allocated into two groups after baseline examination. Group 1 will receive class-integrated DVSS at baseline and then weekly class-integrated social story reinforcement sessions at the first two months, whereas Group 2 will receive 8 weekly social stories reinforcement on an unrelated topic. Both groups will be examined at 3, 6, 12 and 18 months with conventional non-pharmacological behavioural management techniques (CNPBMT). The outcome domains to be evaluated include the time required for the ASD preschool children to complete a compreheisve dental exams, their cooperativeness and anxiety levels during the dental examination, and cost benefits when class-integrated social stories were used with CNPBMT, versus CNPBMT alone.

The knowledge generated can be translated into practice, addressing the current dental barriers and improving patient care among ASD children.

DETAILED DESCRIPTION:
Social story is a training method constituting of short stories to convey information in a step-by-step manner, so that ASD children can understand what to expect and how to behave in different situations in daily lives. Social stories have been implemented to introduce dentistry and improve oral hygiene to individuals diagnosed with ASD with promising results. However, the certainty of evidence for its effectiveness in reducing dental fear during dental visit was low as the results were derived from small-scaled non-randomized controlled studies.

Interventions The intervention group will receive a validated social story ECOHC and reinforcement sessions after baseline recruitment. The control group will not receive any social story or reinforcement session throughout the study period. The randomisation ratio is 1:1.

The developed and validated social story will be distributed to the participants in the intervention group. The same research assistant will visit their SCCCs 8 times to provide weekly class-integrated social story reinforcement sessions at 1-2 months, then the class-integrated social story ECOHC reinforcement will be discontinued. The visiting research assistant will receive training from the team's clinical psychologist, speech-and-hearing therapist, and occupational therapist for the reinforcement sessions.

Oral examinations and NPBBMT for intervention and control groups All children in both groups will receive dental examinations at their respective SCCCs at 3, 6, 12, 18 months. Kindergarten tables lined with mattress and pillows will be set up, and children will be asked to lie supine for oral visual examination using a blunt probe and a disposable front-surface dental mirror attached to light-emitting diode for intra-oral illumination with a disposable plastic sleeve. All examinations will be performed by one single dentist wearing Personal Protective Equipment implementing a standardised protocol of conventional non-pharmacological basic behavioural management techniques (CNPBMT), The time required from the participants being called for examination to completion of the examination will be recorded. If the children continue to refuse to open their mouths and cooperate within the 20-minute appointment time with the standardised CNPBMT employed, no further attempt will be made to perform the examination.

Visible plaque index (VPI) will be first used to assess the baseline oral hygiene level (Ainamo & Bay, 1975). Caries status will be assessed by two parameters: caries diagnostic criteria recommended by WHO (2013), and the modified International Caries Detection and Assessment System (ICDAS). All tooth surfaces will be first wiped clean and dried using a clean gauze and cotton swab before visual inspection of caries. Basic dental charting will be performed, and the overall primary dentition will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Preschool children will be eligible if they have been diagnosed with ASD, following signed parental consent and completion of the questionnaire.
* The proposed study will target Hong Kong preschool children diagnosed with ASD
* Have their full primary dentition erupted
* Able to understand and benefit from social stories (Gray, 2000).

Exclusion Criteria:

* ASD children who have visual or hearing impairments
* Whose parents who cannot read Chinese will be excluded.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The mean appointment time required for the ASD children to complete each proportion of the comprehensive dental examinations | at 3, 6, 12 and 18 months.
  Time required to examine for oral hygiene and dental caries

SECONDARY OUTCOMES:
The proportion of children being cooperative during comprehensive dental examination | at 3, 6, 12 and 18 months.
  Evaluated by Frankl behavioural rating scale (FS) (Frankl, Shiere, & Fogels, 1962). The proportion of children achieving Frankl scale of 3 or 4.
The proportion of children achieving total cooperation during comprehensive dental examination | at 3, 6, 12 and 18 months.
  Evaluated by Venham behavioural rating scale (VS) (Venham et al., 1980). The proportion of children scoring "0" on VS score, i.e. total cooperation
The mean percentage of comprehensive dental examination for oral hygiene and dental caries completed by ASD children within a 20-minute dental appointment time | at 3, 6, 12 and 18 months.
  The dental examination is subdivided into examination of (i) oral hygiene and (ii) dental caries. For oral hygiene, the number of index tooth surfaces that can be examined is recorded divided by 12 index surfaces. Whereas for dental caries, the number of teeth and surfaces that can be viewed and assessed for decay will be divided by 20 primary teeth and 100 surfaces. The mean percentage of the two groups in oral hygiene and dental caries assessment will be compared.
Cost | at 3, 6, 12 and 18 months.
  The overall cost (CCISS) of implementing the class-integrated social stories will be calculated with a bottom-up estimation, including the production cost of the social stories, training cost and implementation cost (CI) with the reinforcement sessions. The implementation cost (CI) is estimated by multiplying the number and duration of the reinforcement sessions with salary of the research assistant (SRA).
Benefits | at 3, 6, 12 and 18 months.
  Assuming that when the ASD children cannot complete over 80% of the comprehensive examination, at least one additional dental appointment has to be rescheduled. At each examination timepoint (3, 6, 12, 18 months), the comparative benefits include (1) the cost savings for an additional appointment, calculated by multiplying the proportion of children who cannot complete 80% of the comprehensive examination by the duration of each additional appointment (20 minutes) along with the wages of the dentist and chairside assistant, as well as adding the material cost; (2) cost savings resulting from a reduction in the average appointment time, calculated by multiplying the mean reduction in time by the combined salaries of the dentist and chairside assistant. As social stories reinforcement and dental examinations will be conducted during class in SCCCs, indirect cost and benefits from the carers' perspective for carers of ASD children will not be considered in this CBA.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on request from the PI. The data are not publicly available as the containing information could compromise the privacy of research participants.